CLINICAL TRIAL: NCT01344512
Title: Population Pharmacokinetics Of Ceftazidime, Ciprofloxacin And Voriconazole In Paediatric Young Patients (< 12 Years Old)
Brief Title: Population Pharmacokinetics of Anti-infectious Drugs in Children
Acronym: PHARMA-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/36
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Pediatrics; Ceftazidime; Ciprofloxacin; Voriconazole
Keywords: Pharmacokinetic; Population; Children; Ceftazidime; Ciprofloxacin; Voriconazole; Pediatric
MeSH Terms: interventions — Ceftazidime; Ciprofloxacin; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients treated with Ceftazidime (Experimental)
  Interventions: Drug: Ceftazidime
- Patients treated with Ciprofloxacin (Experimental)
  Interventions: Drug: Ciprofloxacin
- Patients treated with Voriconazole (Experimental)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Ceftazidime — Bloods sampling on patient treated with Ceftazidime between 48 hours and 4 days after beginning of treatment.
  Arms: Patients treated with Ceftazidime
Drug: Ciprofloxacin — Bloods sampling on patient treated with Ciprofloxacin between 48 hours and 4 days after beginning of treatment.
  Arms: Patients treated with Ciprofloxacin
Drug: Voriconazole — Bloods sampling on patient treated with Voriconazole between 48 hours and 4 days after beginning of treatment.
  Arms: Patients treated with Voriconazole

SUMMARY:
The Pharm A project is a French national collaborative project aiming to determine the population pharmacokinetics of ceftazidime, ciprofloxacin, and voriconazole in paediatric patients aged one month to five years.

DETAILED DESCRIPTION:
The licensing process was introduced in order to ensure that medicines are safe, effective and of high quality. However, over 50% of children admitted to hospital in France and Europe will receive an unlicensed or off-label medicine. This occurs for most drugs in children less than 6 years of age. They represent a particularly vulnerable subgroup of the paediatric population.

There are major practical and ethical issues in relation to studying medicines in paediatric patients aged 5 years or less.

* They represent only a small part of the population as compared to older children and adults, and the variation of specific types of diseases in this young subpopulation is higher than in the paediatric counterpart. There are major differences in drug disposition in the different age groups.
* There is a need for suitable methodological approaches for clinical trials
* There are major ethical issues It is essential, therefore, to recruit children from various regions in France in order to obtain a critical sample size of sufficient magnitude and to conduct scientific sound studies. This will be achieved by performing Pharm A, a population pharmacokinetic study of three different anti infectious agents (ceftazidime, ciprofloxacin, voriconazole) and identify covariates including pharmacogenetic biomarkers that explain pharmacokinetic variability.

After parental informed consent, sampling strategy will be randomized depending on the drug and the age group (2 samples in patients below 2 years and 3 samples in patients from 2 to 5 years).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 28 days to 11 years (< 12 years)
* Receiving one of the following drugs for therapeutic reasons : ceftazidime, ciprofloxacin, voriconazole
* Representative for the clinician, a condition requiring the use of these molecules
* Informed consent signed by the two parents or legal representative
* Child affiliated to the national social security system

Exclusion Criteria:

Not Applicable

Ages: 28 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Population pharmacokinetic parameters and factors explaining variability | Between 2 and 4 days after the begining of the treatment
  Population Pharmacokinetic Parameters and variability factors (Sex, Age, Genetic factors...) for ceftazidime, ciprofloxacin and voriconazole.
  According to the age of participants, 2 or 3 bloods sampling will be take between 2 and 4 days after the beginning of the treatment.

SECONDARY OUTCOMES:
Covariability factors explaining the variability (age, biological data, pharmacokinetics factors, associated treatments...) | Between 2 and 4 days after the beginning of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Bui, Dr, Principal Investigator — University Hospital Bordeaux, France
Locations (14):
- France (14):
  - CHU de Bordeaux, Hôpital Pellegrin, Bordeaux
  - Hospices Civils de Lyon, Bron
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU Lille, Lille
  - AP-HM, Hôpital La Timone, Marseille
  - CHU Montpellier, Montpellier
  - APHP - Hôpital NEcker, Paris
  - AP-HP - Hôpital Robert Debré, Paris
  - CHU Poitiers, Poitiers
  - CHU Rouen, Rouen
  - CHU Toulouse, Toulouse
  - CHU tours, Tours

REFERENCES:
- [Derived] Bui S, Facchin A, Ha P, Bouchet S, Leroux S, Nacka F, Fayon M, Jacqz-Aigrain E. Population pharmacokinetics of ceftazidime in critically ill children: impact of cystic fibrosis. J Antimicrob Chemother. 2020 Aug 1;75(8):2232-2239. doi: 10.1093/jac/dkaa170. PMID 32457995